CLINICAL TRIAL: NCT02536573
Title: Prospective, Randomized Study to Evaluate Total Hip Arthroplasty With and Without Radlink Surgical Positioning Software
Brief Title: Study of Total Hip Arthroplasty Using Radlink Surgical Positioning Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anderson Orthopaedic Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AORI 2015-0101
Record Dates: First submitted 2015-08-24; First posted 2015-09-01 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Total Hip Replacement
Keywords: Total hip replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Intraoperative fluoroscopy of the hip is used to visually estimate the acetabular cup angle and make any necessary adjustments.
- Radlink Surgical Positioning System (Experimental): Fluoroscopic image of the hip joint is imported into the Radlink Surgical Positioning software. The software calculates a target cup position using bony landmarks, and the surgeon matches the cup to the target.
  Interventions: Other: Radlink Surgical Positioning Software

INTERVENTIONS:
Other: Radlink Surgical Positioning Software
  Arms: Radlink Surgical Positioning System

SUMMARY:
This is a prospective, randomized study of total hip arthroplasty with and without the use of Radlink surgical positioning software. The investigators are interested in discovering whether the use of the Radlink software will provide more accurate acetabular cup position when compared with surgeon estimates based on visual inspection of fluoroscopic images.

ELIGIBILITY:
Inclusion Criteria:

* Total hip arthroplasty

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Radiographic cup abduction angle | 4 month postoperative
  Angle of acetabular component in coronal plane measured on x-ray
Radiographic cup anteversion angle | 4 month postoperative
  Angle of acetabular component in sagittal plane measured on x-ray

SECONDARY OUTCOMES:
Variance of cup angles measured on x-ray | 4 month postoperative
  Statistical homogeneity of angles and how spread out the data is.

CONTACTS AND LOCATIONS:
Overall Officials: William G Hamilton, MD, Principal Investigator — AORI (Anderson Orthopaedic Research Institute)